CLINICAL TRIAL: NCT01151527
Title: Genetics, Genomics, and Proteomics of Idiopathic Interstitial Pneumonias: Identification of Susceptibility Genes, Biomarkers, and Molecular Phenotyping
Brief Title: Peripheral Blood Biomarkers in Idiopathic Interstitial Pneumonias
Status: Terminated | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Jewish Health (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00022485; R01HL097163-01 (NIH); RC1HL099571 (NIH)
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2010-06

CONDITIONS: Idiopathic Interstitial Pneumonias
MeSH Terms: conditions — Idiopathic Interstitial Pneumonias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tubes of blood will be drawn from the subject to extract RNA and DNA for laboratory purposes.
  Lung biopsy tissue (pathology slides) may be requested for specimen processing.
  Also Bronchoscopy fluid may be requested.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sporadic (idiopathic) or familial interstitial pneumonia: We are recruiting patients with Idiopathic Pulmonary Fibrosis and other types of Idiopathic Interstitial Pneumonias that occur sporadically or familial (2 or more affected individuals in a family). Participation can be done by mail or visiting Duke University Medical Center (Durham, NC)or National Jewish Health (Denver, CO).

SUMMARY:
We hypothesize that a peripheral blood biomarker or biological signature (gene or protein expression pattern) of idiopathic interstitial pneumonias (IIPs) will simplify and improve the accuracy of diagnosis of IIP and diagnose individuals at an earlier, more treatable, stage of their disease.

DETAILED DESCRIPTION:
The Broad Challenge Area addressed in this proposal is (03) Biomarker Discovery and Validation, and the Specific Challenge Topic is 03-HL-101 (Identify and validate clinically relevant, quantifiable biomarkers of diagnostic and therapeutic responses for blood, vascular, cardiac, and respiratory tract dysfunction). Idiopathic interstitial pneumonia (IIP) is a lung disease(s) that primarily affects the elderly, but is present in all age groups. IIP causes respiratory insufficiency and is often fatal. In about half of the patients, the diagnosis requires an invasive lung biopsy which can cause complications, and is not always accurate.

The current diagnostic tools for IIP are inadequate. In addition to inaccurate diagnosis, they are very costly, and often result in delayed diagnosis and treatment. The challenge(s) we intend to address in this proposal is to improve the accurate and early diagnosis of idiopathic interstitial lung pneumonia (IIP), and to improve the ability to differentiate the subtypes of idiopathic interstitial pneumonias (IIPs) by developing peripheral blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Sporadic cases of Idiopathic Pulmonary Fibrosis and other types of Idiopathic Interstitial Pneumonias.
* Family members ( with or without clinical disease) with a family history of pulmonary fibrosis.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are recruiting patients with Idiopathic Pulmonary Fibrosis and other types of Idiopathic Interstitial Pneumonias that occur sporadically or familial (2 or more affected individuals in a family).
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2010-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Steele, MD, Principal Investigator — Duke University; David A Schwartz, MD, Principal Investigator — National Jewish Health
Locations (2):
- United States (2):
  - National Jewish Health, Denver, Colorado
  - Duke University Medical Center, Durham, North Carolina